CLINICAL TRIAL: NCT05973643
Title: Study by 1H NMR of the Variations of the Metabolome During the Course of Electroconvulsive Therapy in Patients With Major Depressive Episode
Brief Title: Metabolomics During ElectroConvulsivoTherapy
Acronym: METECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A00548-37
Record Dates: First submitted 2023-07-17; First posted 2023-08-03 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Episode; ECT
Keywords: 1HNMR; Electroconvulsive Therapy; Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Electroconvulsive Therapy

STUDY DESIGN:
Intervention Model Description: simple-blind, any adult patient presenting a characterized depressive episode in the context of unipolar major depressive disorder or bipolar disorder who consents and requires an ECT treatment. study including 50 patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electroconvulsive therapy (Other): simple-blind, any adult patient presenting a characterized depressive episode in the context of unipolar major depressive disorder or bipolar disorder who consents and requires an ECT treatment. study including 50 patients.
  Interventions: Other: Electroconvulsive therapy

INTERVENTIONS:
Other: Electroconvulsive therapy — Electroconvulsive therapy is administered through electrodes positioned bilaterally (bitemporal) or unilaterally (or fronto-temporal) on the frontotemporal region under anesthesia.
  The stimulation dose is determined by titration method, during the first ECT session. An ECT cure corresponding from 12 to 20 sessions of ECT. Patients will receive 2 sessions a week.
  Blood samples will be done during the anesthesia process.

SUMMARY:
Investigators will measure the variation of blood Metabolome through 1H NMR at several time points during the course of electroconvulsivetherapy in patients with a major depressive episode. Patients with a major depressive disorder or a bipolar disorder and a current major depressive episode will be included in this study. Investigators hypothesized that Metabolome could be a source to predict response during ECT and to help understanding underlying biological mechanisms.

DETAILED DESCRIPTION:
Biological signatures of blood metabolome will be measure before and after the first session of electroconvulsivetherapy, and during the course, before the 6th, 12th and the last sessions. Proton Nuclear Magnetic Resonance spectroscopy will be used to measure metabolites in blood sample. In parallel, at each time point, depression severity (MADRS and BDI), Perceived severity (CGI), global functioning (EGF), convulsive characteristics and cognitive tolerance (MOCA) will be measure, at each time point.

The aim of this study is to determine whether 1HNMR could help to understanding metabolic ways and predict response to ECT in patients with a current Major Depressive Episode (MDE) in Major Depressive Disorder (MDD) and in Bipolar Disorder (BD).

To date, scientific community knows that ECT is a safety and efficacy treatment in MDE particularly resistant or severe, but scientific community knows little about its mechanism of action.

The investigators hypothesize that 1HNMR could help to go further.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive episode according to DSM-5 criteria
* Diagnosis of major depressive disorder or bipolar disorder
* MADRS score >22
* having given written, free and informed consent
* without protective measures
* resistance criterion defined as failure of 2 antidepressants at an effective dose for a minimum of 6 weeks
* current major depressive episode according to DSM-5 criteria with indication of treatment by ECT cure

Exclusion Criteria - Cannot be included in the study, people:

* whose consent is not admissible or who refuse to participate in the study
* deprived of liberty by judicial or administrative decision
* For which there is a particular risk contraindicating the cure of ECT
* Suffering from schizophrenia spectrum disorders or persistent delusional disorder as described by DSM-5 Criterion D for Major Depressive Disorder
* suffering from neurological disorders (such as patients suffering from multiple sclerosis, epilepsy, encephalitis, etc.) and/or neurodegenerative disorders (such as Parkinson's disease, Alzheimer's disease or related diseases, etc.) as described by criterion C of the major depressive disorder listed in the DSM-5
* suffering from an acute or chronic systemic inflammatory disease requiring specific treatment with immunomodulators or suppressors. As well as any recurrent inflammatory disease requiring specific management, and which may lead to a differential diagnosis of the characterized depressive episode as described by criterion C listed in the DSM-5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Value the metabolic profile difference between the baseline and before the 6th session of ECT by blood metabolomics through 1HNMR | up to 3 weeks
  identify variations in the metabolome by measuring the metabolome in the blood of patients treated for depressive episodes or bipolar disorder by identifying the metabolic profiles associated with the medical response to ECT between the Baseline and before the sixth ECT session.

SECONDARY OUTCOMES:
Measure the biological effect of one ECT session on the blood metabolome | through first ECT session, an average of 1 week
  Comparison of quantitative and qualitative measurements of metabolites and metabolic signatures obtained by 1HNMR between baseline and the first ECT by observing either a clinical response or a clinical remission by discriminating remitters and no remitters patients.
Compare the biological effect measured between the baseline and before the 1st, 6th and 12th session of ECT | through study completion, up to 6 weeks
  Comparison of quantitative and qualitative measurements of metabolites and metabolic signatures obtained by 1HNMR between baseline and the first ECT by observing either a clinical response or a clinical remission by discriminating remitters and no remitters patients. The clinical response is defined by the decrease of 50% on the MADRS scale. The clinical remission is defined by a score less than or equal to 10 on the MADRS scale.
Measure the variations of the metabolic signature according to the clinical response during the ECT treatment | up to 10 weeks
  Comparison of quantitative and qualitative measures of metabolites taken separately and metabolic signatures obtained by 1H NMR according to the clinical response on the MADRS scale (the overall score thus ranges from 0 to 60) throughout the course of ECT. The clinical response is defined by the decrease of 50% on the MADRS scale. The clinical remission is defined by a score less than or equal to 10 on the MADRS scale.
Look for a metabolic signature to discriminate between responder and non-responder patients before the 6 ECT sessions (i.e. the day of the 6th) | through the sixth session, up 3 weeks
  Comparison of metabolic signatures obtained by very high field NMR between responder and non-responder patients before the 6th ECT session (V2)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier le Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aberg-Wistedt A, Martensson B, Bertilsson L, Malmgren R. Electroconvulsive Therapy Effects on Cerebrospinal Fluid Monoamine Metabolites and Platelet Serotonin Uptake In Melancholia. Convuls Ther. 1986;2(2):91-98. PMID 11940851
- [Result] Abrams R, Essman WB, Taylor MA, Fink M. Concentration of 5-hydroxyindoleacetic acid, homovanillic acid, and tryptophan in the cerebrospinal fluid of depressed patients before and after ECT. Biol Psychiatry. 1976 Feb;11(1):85-90. PMID 1260078
- [Result] van Diermen L, van den Ameele S, Kamperman AM, Sabbe BCG, Vermeulen T, Schrijvers D, Birkenhager TK. Prediction of electroconvulsive therapy response and remission in major depression: meta-analysis. Br J Psychiatry. 2018 Feb;212(2):71-80. doi: 10.1192/bjp.2017.28. PMID 29436330
- [Result] Yatham LN, Kennedy SH, Parikh SV, Schaffer A, Bond DJ, Frey BN, Sharma V, Goldstein BI, Rej S, Beaulieu S, Alda M, MacQueen G, Milev RV, Ravindran A, O'Donovan C, McIntosh D, Lam RW, Vazquez G, Kapczinski F, McIntyre RS, Kozicky J, Kanba S, Lafer B, Suppes T, Calabrese JR, Vieta E, Malhi G, Post RM, Berk M. Canadian Network for Mood and Anxiety Treatments (CANMAT) and International Society for Bipolar Disorders (ISBD) 2018 guidelines for the management of patients with bipolar disorder. Bipolar Disord. 2018 Mar;20(2):97-170. doi: 10.1111/bdi.12609. Epub 2018 Mar 14. PMID 29536616